CLINICAL TRIAL: NCT03187028
Title: Diet and Exercise After Pancreatic Cancer: Clinical and Functional Outcomes (Non Canonical WNT Signaling in Colorectal Cancer)
Brief Title: Diet and Exercise After Pancreatic Cancer
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: F141218007
Record Dates: First submitted 2017-05-24; First posted 2017-06-14 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: Cancer of Pancreas; Neoplasms, Pancreatic; Pancreas Cancer; Pancreas Neoplasms; Cancer of the Pancreas; Pancreatic Cancer; Foregut Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet only (Active Comparator): Diet counseling will be delivered using visual communication (e.g., Skype). Participants will be provided a computer tablet for the intervention with participants randomized to receive diet counseling.
  Interventions: Behavioral: Diet Only
- Diet + Exercise (Experimental): Diet and exercise counseling will be delivered using visual communication (e.g., Skype). Participants will be provided a computer tablet for the intervention with participants randomized to receive diet and exercise counseling also receiving a fitness bracelet to facilitate counseling by the certified Cancer Exercise Trainer.
  Interventions: Behavioral: Diet + Exercise

INTERVENTIONS:
Behavioral: Diet Only — Diet counseling will be delivered using visual communication (e.g., Skype). Participants will be provided a computer tablet for the intervention with participants randomized to receive diet counseling.
  Arms: Diet only
Behavioral: Diet + Exercise — Diet and exercise counseling will be delivered using visual communication (e.g., Skype). Participants will be provided a computer tablet for the intervention with participants randomized to receive diet and exercise counseling.
  Arms: Diet + Exercise

SUMMARY:
Determine feasibility of a randomized controlled trial (RCT) in pancreatic (& other foregut) cancer patients comparing the effects of diet alone vs. diet+exercise on functional and clinical outcomes.

DETAILED DESCRIPTION:
Foregut cancers such as pancreatic cancer cause significant side effects and poorer health-related quality of life (QOL), as well as a 5-year survival rate of only 6%. Importantly, the reduction in physical functioning caused by this cancer and its therapies is associated with higher mortality risk. Although multiple studies in more prevalent cancer types support exercise benefits (e.g., improved physical functioning), data cannot be generalized from one cancer type to another. Little is known about exercise feasibility and benefits in pancreatic (& other foregut) cancer patients, and no data regarding potential mechanistic outcomes that may explain the link between poor physical performance status and cancer survival have been reported. We will enroll 20 patients with pancreatic adenocarcinoma (or other foregut cancer) who are expected to undergo surgical resection or who are within 3 years of surgical resection, in a pilot project involving a 6-month home-based lifestyle intervention (diet along versus diet+exercise). Research assessments will be done pre-surgery (if applicable), post-surgery (and prior to starting the intervention), 3 months, and 6 months post-surgery. Intervention counseling will be delivered using visual communication (e.g., Skype). Participants will be provided a computer tablet for the intervention with participants randomized to receive exercise counseling also receiving a fitness bracelet to facilitate counseling by the certified Cancer Exercise Trainer. Our primary study aim is to determine feasibility of a randomized controlled trial (RCT) in pancreatic cancer patients comparing the effects of diet alone with diet+exercise on pancreatic cancer-related functional and disease outcomes; feasibility measures include recruitment, retention, intervention adherence, assessment completion, adverse events, and participant satisfaction. Our secondary study aim is to determine the effect of diet+exercise compared with diet alone on physical functioning and QOL. Also, we will draw and store blood samples so that additional funds can be requested to test intervention effects on biomarkers of cancer risk (e.g., tumor immunity, inflammatory cytokines, etc.). The goal of the study is to advance the exercise oncology field into an understudied cancer type and develop an intervention that will improve the survivorship care of pancreatic cancer patients through distance-delivered counseling methods.

ELIGIBILITY:
Inclusion Criteria:

* adult 18 years of age or older with resectable foregut cancer for whom surgery is planned (includes "borderline resectable" if deemed appropriate by surgical investigators) or has occurred within the past 3 years
* English speaking
* Eastern Cooperative Technology Group (ECOG) performance status of 0,1 or 2.
* able to ambulate without assistance
* able to obtain medical clearance

Exclusion Criteria:

* foregut cancer recurrence
* dementia or organic brain syndrome
* severe emotional distress
* medical, psychological or social characteristic that would interfere with the ability to fully participate in program activities and assessments
* another diagnosis of cancer in the past 5 years (not including skin or cervical cancer in situ).
* oncologist refuses to allow screening for possible study participation
* current participation in another exercise trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Baseline
  Number of participants excluded or not agreeing to participate
Feasibility - Adherence to study protocol activities | Throughout 6 month study period
  Feasibility measure (e.g. percent of assessments completed, percent of counseling sessions completed, etc.)
Feasibility - Attrition rates | Throughout 6 month study period
  Number of participants who dropout or are withdrawn
Feasibility - Adverse events | Throughout 6 month study period
  Recorded by staff
Feasibility - Participant satisfaction | At conclusion of 6 month study period
  Survey

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) performance status | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Preliminary effect size
Quality of life (assessed using the Functional Assessment of Cancer Therapy index) | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Preliminary effect size
Objective physical functioning | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Preliminary effect size
CA 19-9 (tumor markers) | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Exploratory data related to within and between group (diet and diet+exercise) differences
Completion of pancreatic cancer treatment | At conclusion of 6 month study
  Exploratory data related to within and between group (diet and diet+exercise) differences
Survival rates | At conclusion of 6 month study
  Exploratory data related to within and between group (diet and diet+exercise) differences
Pancreatic cancer recurrence rates | At conclusion of 6 month study
  Exploratory data related to within and between group (diet and diet+exercise) differences
Prognostic blood cytokine biomarkers | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Exploratory data related to within and between group (diet and diet+exercise) differences
Prognostic blood tumor immunity biomarkers | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Exploratory data related to within and between group (diet and diet+exercise) differences
Wearable activity monitor (weekly minutes of physical activity) | At 4 timepoints during the 6 month study (pre-surgery if applicable, post-surgery/prior to starting the intervention, 3 months and 6 months)
  Exploratory data related to within and between group (diet and diet+exercise) differences

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided